CLINICAL TRIAL: NCT06505577
Title: Concordance Between Preoperative Assessments and Pathologic Size Measurements in Breast Cancer: a Prospective Observational Study
Brief Title: Preoperative vs. Pathologic Size in Breast Cancer: A Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Incheon St.Mary's Hospital (Other)
Collaborators: Yonsei University (Other)
Responsible Party: Principal Investigator, Young-Joon Kang, Assistant Professor, Incheon St.Mary's Hospital
Other Study IDs: PREPARE-01
Record Dates: First submitted 2024-07-04; First posted 2024-07-17 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Mastectomy; Breast Neoplasm Malignant Primary
Keywords: Breast cancer; Mastectomy; Ductal carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Breast cancer surgery group: This cohort includes all patients undergoing breast cancer surgery who are enrolled in the study.
  Interventions: Other: No additional intervention

INTERVENTIONS:
Other: No additional intervention — All patients are scheduled to undergo standard breast surgery as part of their routine clinical care. No additional interventions are administered specifically for this study.

SUMMARY:
Breast cancer, the most prevalent malignancy among women globally, is increasing in incidence. While non-metastatic breast cancer requires surgery, determining the optimal extent of resection remains challenging. Inadequate resection margins necessitate reoperation, leading to increased psychological stress, costs, and potentially compromised cosmetic outcomes and prognosis.

Accurate preoperative assessment of resection extent is crucial and involves various factors, including imaging studies, physical examinations, tumor molecular subtypes, and intraductal carcinoma components. This prospective observational study aims to identify and integrate multiple predictive factors to enhance surgical planning and minimize reoperation rates in breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is the most prevalent malignancy among women globally, leading to surgical interventions for non-metastatic cases. While breast cancer generally has a favorable prognosis, achieving negative resection margins at initial surgery is crucial for optimal outcomes. The challenge associated with accurately predicting the extent of resection preoperatively, as failure to secure clear margins may necessitate further resection or total mastectomy, resulting in increased psychological stress, higher healthcare costs, compromised cosmetic results, and potential negative impacts on long-term prognosis and quality of life. Many factors contribute to predicting the optimal resection extent, including imaging studies, physical examination findings, tumor molecular subtypes, presence and extent of intraductal carcinoma components, etc. Despite the availability of these predictive factors, their integration and practical application in clinical decision-making remain challenging. This prospective observational study aims to address this gap by analyzing the interplay of these factors in real-world clinical settings, with the primary objective of deriving an integrated predictive model to guide surgeons in determining the optimal extent of resection preoperatively.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥ 19 years old) diagnosed with breast cancer (invasive and in situ).

Patients scheduled for surgical resection of the tumor Availability of both preoperative tumor size assessments and pathologic measurements post-surgery

Exclusion Criteria:

Patients with recurrent breast cancer Inflammatory breast cancer Patients who did not undergo surgery Patients whose preoperative tumor size data is not available or deficient for analyzing

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be enrolled from patients at Incheon Saint Mary's Hospital, a 1000-bed tertiary academic medical center located in Incheon, South Korea.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Concordance rate by the intraclass correlation coefficient Factors associated with discrepancies | Within 30 days after surgery
  To assess the concordance between preoperative tumor size assessments made by surgeons and the actual tumor size determined by pathologic analysis following surgical resection in patients with breast cancer.
  * Using the scale of Landis and Koch according to the intraclass correlation coefficient.
  * With/without MRI status. To identify and evaluate factors associated with discrepancies between preoperative assessments and pathologic measurements.

SECONDARY OUTCOMES:
Concordance rate by size discordance (5mm) To evaluate the concordance between preoperative tumor size assessments and pathologic measurements in the subgroup of patients with ductal carcinoma in situ (DCIS) | Within 30 days after surgery
  To assess the concordance between preoperative tumor size assessments made by surgeons and the actual tumor size determined by pathologic analysis following surgical resection in patients with breast cancer. A difference of 5mm or more between preoperative and pathologic measurements is defined as discordance.
Concordance rate and discrepancy factor in ductal carcinoma in situ (DCIS) subgroup | Within 30 days after surgery
  To evaluate the concordance between preoperative tumor size assessments and pathologic measurements in the subgroup of patients with ductal carcinoma in situ (DCIS).
Concordance rate and discrepancy factor in neoadjuvant systemic therapy subgroup | Within 30 days after surgery
  To assess the concordance between preoperative tumor size assessments and pathologic measurements in the subgroup of patients who received neoadjuvant systemic therapy
Proportion of surgical method change: rates of unnecessary total mastectomy | Within 30 days after surgery
  To determine the rate of change in surgical method (e.g., from lumpectomy to mastectomy, nipple-sparing to skin-sparing, or vice versa) based on discrepancies between preoperative tumor size assessments and pathologic measurements. This involves collecting the initial surgical method plan from the surgeon before the surgery and, after confirming the pathological size post-surgery, collecting the final surgical method deemed feasible for the patient from the surgeon.
Factors requiring MRI: factors associated with size discrepancy between MRI and mammography (with/without Breast ultrasonography) | Within 30 days after surgery
  To determine the associated factors contributing to size discrepancies between mammography (with or without breast ultrasonography) and MRI. For analyzing the clinical factors that necessitate the use of MRI to predict the pathologic tumor size.
Rate of recurrence within 1-year after breast surgery | Within 1 year after enroll
  The proportion of patients who develop new malignant lesions during the follow-up period within 1 year after breast surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Incheon St. Mary's Hospital, Incheon, South Korea